CLINICAL TRIAL: NCT01579214
Title: Cell Phone Messaging to Improve Communication of Critical Laboratory Results to Patients in Rural Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other); Fogarty International Center of the National Institute of Health (NIH); Harvard University (Other)
Responsible Party: Principal Investigator, Mark Siedner, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011P001538; R24TW007988 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: HIV; Tuberculosis
Keywords: HIV; Africa south of the sahara; Knowledge of results; Communication barriers; Cellular Phones
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental design study with two periods of study. The pre-intervention period serves as the control group. During the intervention period, participants received one of three message types to be informed of their test results: 1) a standard message informing their abnormal result, 2) the standard message protected by a PIN number code, and 3) a coded texted message "ABCDEFG."
  For our a priori hypotheses about the effect of receiving an SMS message on outcomes, we compared results for participants in the pre-intervention period with all those in the post-intervention period. This was a non-randomized intervention.
  For our primary outcome (time to ART initiation) we assessed all participants with abnormal CD4 count results who were ART-naive at study enrollment. For our secondary outcome (time to clinic return) we looked at all study participants with abnormal CD4 counts.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Text Message (Active Comparator): Participants in the intervention period (September 2012 - November 2013) received daily short message service (SMS) messages for up to seven days with messages reporting an abnormal result
  Interventions: Other: Cellular Phone Text Messages
- Pre-Intervention (No Intervention): Participants enrolled in the pre-intervention period (January - August 2012) served as a control group.

INTERVENTIONS:
Other: Cellular Phone Text Messages — Cellular phone text message formats to be sent to participants after abnormal laboratory results to communicate information and request early return to clinic.
  Arms: Direct Text Message

SUMMARY:
The investigators will study the efficacy of a novel cellular phone messaging system to communicate health information and facilitate early return to clinic after abnormal laboratory results in rural Uganda.

DETAILED DESCRIPTION:
Among the challenges that complicate optimal health care delivery in rural settings is lack of communication between care providers and patients. Communication of abnormal laboratory results represents a particular challenge. Laboratory and other test results are often not reported until repeat visits weeks to months later. In the case of treatment failure, severe treatment complications, or evidence of opportunistic infection, such reporting delays likely result in adverse outcomes and potentially compromise future treatment options. The investigators propose to evaluate a novel strategy of communication using SMS text messaging to facilitate patient return to an HIV clinic in Uganda after critical laboratory results.

The investigators will consent and enroll participants at the time of laboratory testing for cluster of differentiation 4 (CD4) count, viral loads, acid fast bacteria smears of sputum, among others. Those with abnormal results will be randomized to various messaging formats and receive text messages requesting a prompt return to clinic. For outcomes, the investigators will measure successful receipt and comprehension of messages, as well as proportion returning within 14 days of the abnormal laboratory test.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Active in care at Mbarara Regional Referral Hospital HIV Clinic
* Undergoing laboratory testing
* Self-reported cell phone access
* Agrees to participation and gives informed consent

Exclusion Criteria:

* Age < 18
* Resides outside great Mbarara area (Mbarara, Isingiro, Kyruhuura, Ibanda, or Ntungamo districts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Siedner, MD MPH, Study Director — Massachusetts General Hospital; Bosco Bwana, MD, Principal Investigator — Mbarara University of Science and Technology; David R Bangsberg, MD MPH, Principal Investigator — Massachusetts General Hospital Center for Global Health; Jessica Haberer, MD MS, Principal Investigator — Massachusetts General Hospital Center for Global Health
Locations (1):
- ISS Clinic, Mbarara Regional Referral Hospital, Mbarara, Uganda

REFERENCES:
- [Result] Siedner MJ, Haberer JE, Bwana MB, Ware NC, Bangsberg DR. High acceptability for cell phone text messages to improve communication of laboratory results with HIV-infected patients in rural Uganda: a cross-sectional survey study. BMC Med Inform Decis Mak. 2012 Jun 21;12:56. doi: 10.1186/1472-6947-12-56. PMID 22720901
- [Result] Siedner MJ, Santorino D, Lankowski AJ, Kanyesigye M, Bwana MB, Haberer JE, Bangsberg DR. A combination SMS and transportation reimbursement intervention to improve HIV care following abnormal CD4 test results in rural Uganda: a prospective observational cohort study. BMC Med. 2015 Jul 6;13:160. doi: 10.1186/s12916-015-0397-1. PMID 26149722
- [Result] Siedner MJ, Santorino D, Haberer JE, Bangsberg DR. Know your audience: predictors of success for a patient-centered texting app to augment linkage to HIV care in rural Uganda. J Med Internet Res. 2015 Mar 24;17(3):e78. doi: 10.2196/jmir.3859. PMID 25831269

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Intervention Control Group: Participants followed prior to SMS intervention as a negative control group.
- Intervention Group: Received a text message stating laboratory results were abnormal and requesting return to clinic.
Period: Overall Study
Arm/Group | Pre-Intervention Control Group | Intervention Group
Started | 45 | 138
Completed | 45 | 138
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the trial were in HIV care and had low CD4 count results requiring a prompt return to clinic as advised by a study clinician.
Groups:
- Pre-Intervention Control Group: Eligible participants from a pre-intervention period (January-August 2012) prior to their receiving SMS messages about their laboratory test results. During the pre-intervention stage, clinicians completed eligibility forms for each participant, including confirmation of access to a cellular phone, district of residence, and selection of the abnormal result threshold for the cluster of differentiation 4 (CD4) test, which would prompt a request for an early return to clinic. Standard clinical forms were completed to collect data on sociodemographic and clinical characteristics. We also collected data on the laboratory result and result date, time from laboratory result to clinic return, and for antiretroviral therapy (ART) naive participants, time to ART initiation.
- Intervention Period: Participants in the intervention period (September 2012 - November 2013) were receive daily short message service (SMS) messages for up to seven days in one of three formats: 1) messages reporting an abnormal result directly, 2) personal identification number-protected messages reporting an abnormal result, or 3) messages reading "ABCDEFG" to confidentially convey an abnormal result.
  For our a priori hypothesis, we aimed to test whether clinical outcomes, i.e. time to clinic return and time to ART initiation, were different in the pre-intervention and intervention period. This was a non-randomized allocation.
  During the intervention period, clinicians used eligibility criteria identical to those used during the pre-intervention period, including selection of an abnormal cluster of differentiation 4 (CD4) count threshold to trigger the SMS and transportation reimbursement intervention.
- Total: Total of all reporting groups
Arm/Group | Pre-Intervention Control Group | Intervention Period | Total
Number analyzed (Participants) | 45 | 138 | 183
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [31 to 44] | 30 [25 to 38] | 32 [26 to 39]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female Gender | 19 | 75 | 94
  Male Gender | 26 | 63 | 89
Region of Enrollment [Count of Participants; unit: Participants]
  Uganda: Mbarara Resident | 32 | 83 | 115
  Uganda: Non-Mbarara Resident | 13 | 55 | 68
Number of Antiretroviral Therapy (ART) Naive Participants [Count of Participants; unit: Participants] | 26 | 110 | 136
Educational Attainment [Count of Participants; unit: Participants]
  <Primary | 3 | 12 | 15
  Any primary | 16 | 71 | 87
  Any secondary | 12 | 37 | 49
  >Secondary | 7 | 18 | 25
  Missing Information | 7 | 0 | 7
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 185 [106 to 262] | 225 [110 to 293] | 215 [106 to 285]
Days from enrollment until laboratory result [Median (Inter-Quartile Range); unit: Days] | 11 [8 to 19] | 10 [8 to 15] | 10 [8 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Participants Initiating Antiretroviral Therapy (ART) Within 28 Days of Abnormal Result
Description: Number of Antiretroviral Therapy (ART) naive participants (subgroup of the sample) who initiated ART within 28 days of receiving abnormal result
Time Frame: 28 days
Population: These are participants who were Antiretroviral Therapy naive, and so analysis of this measurement is using this subgroup only.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention Control Group | Intervention Period
Number analyzed (Participants) | 26 | 110
Participants | 8 | 89

2. Secondary Outcome: Clinic Return Within 28 Days of Abnormal CD4 Count Result
Description: Number of participants who returned to clinic within 28 days of abnormal CD4 count result
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention Control Group | Intervention Period
Number analyzed (Participants) | 45 | 138
Participants | 22 | 128

ADVERSE EVENTS:
Time Frame: Study participants were monitored until the time of clinic return which extended to a maximum of approximately 6 months.
Groups:
- Intervention Period: Participants in the intervention period (September 2012 - November 2013) were randomized to receive daily short message service (SMS) messages for up to seven days in one of three formats: 1) messages reporting an abnormal result directly, 2) personal identification number-protected messages reporting an abnormal result, or 3) messages reading "ABCDEFG" to confidentially convey an abnormal result.
  During the intervention period, clinicians used eligibility criteria identical to those used during the pre-intervention period, including selection of an abnormal cluster of differentiation 4 (CD4) count threshold to trigger the SMS and transportation reimbursement intervention.
Arm/Group | Pre-Intervention Control Group | Intervention Period
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/138
Other Adverse Events (participants affected / at risk) | 0/45 | 0/138

LIMITATIONS AND CAVEATS:
1. Non-randomized allocation for primary analysis
2. Single site study
3. Requires validation in implementation study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No